CLINICAL TRIAL: NCT05336903
Title: Development and Feasibility Testing of an Advanced Practice Physiotherapy Role in Chronic Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Miller, PT, PhD (Other)
Collaborators: University Hospitals Kingston Foundation - Women's Giving Circle (Unknown)
Responsible Party: Sponsor-Investigator, Jordan Miller, PT, PhD, Assistant Professor, School of Rehabilitation Therapy, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REH-782-20
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Feasibility study
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a single-arm feasibility study at the one chronic pain clinic in Kingston, Ontario, Canada. The intervention is the integration of an APP as the first point of contact in this interprofessional setting.
Masking Description: Participants will be invited to participate in the study with an understanding that they will be assigned to either a model of care in which they see the physician or nurse practitioner first or a model of care in which they see a physiotherapist first, even though this is a single arm feasibility study and all participants will be assigned to the APP model of care. This partial masking at the time of consent and initial assessment was determined to be important to provide accurate estimates of feasibility (e.g. consent rate, percentage of consenting participants who see the physiotherapist first who also request to see the physician or nurse practitioner). Due to the nature of the intervention, participants and healthcare providers will not be blinded to the intervention received in this or the fully powered trial. Since the primary outcome measures are self-report measures (ie. the participant is the assessor), the outcome assessor is similarly not planned to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APP-led model of care for chronic pain management (Experimental): The APP-led model of care involves integrating an APP as the first point of contact within an interprofessional chronic pain clinic setting. This is in contrast to the usual physician- or nurse practitioner-led model of care.
  Interventions: Behavioral: APP-led model of care for chronic pain management

INTERVENTIONS:
Behavioral: APP-led model of care for chronic pain management — The APP will provide an assessment using a biopsychosocial approach. The assessment will include:
  * taking a comprehensive history
  * screening for pathologies contributing to the participant's chronic pain
  * a physical assessment
  * screening for comorbid health conditions, using the appropriate screening tools, that require specific care (e.g., depression, addiction, post-traumatic stress)
  * identifying psychosocial risk factors associated with pain and disability
  * evaluating pain severity and interference
  The APP will make recommendations to the participant and the chronic pain clinic health care team based on findings from the comprehensive assessment. These recommendations include, but are not limited to, the need for urgent or emergent referrals, medication management, referral and integration of other health care providers, the need for interventional procedures, or group-based treatment options.

SUMMARY:
The current study is intended to evaluate the feasibility of conducting a future trial to evaluate the effects of implementing an advanced practice physiotherapist (APP) role within a chronic pain clinic setting.

DETAILED DESCRIPTION:
This line of research ultimately seeks to assess the impact of integrating an APP as the first point of contact within interprofessional chronic pain clinics on patient health outcomes, care provided to patients, chronic pain clinic flow, and cost-utility in comparison to usual physician or nurse practitioner-led care.

The primary objectives of the feasibility study are:

1. To determine the feasibility of implementing the trial methods by evaluating participant recruitment rates, retention, and assessment completion at each of four follow-up time-points over a 12-month period.
2. To determine the feasibility of implementing the new APP model of care by monitoring the care provided and treatment fidelity.
3. To explore the perspectives of participants and health care providers related to the acceptability of the APP role; barriers, facilitators, and strategies for refining implementation; and perceived impact on clinic processes and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic musculoskeletal pain (pain > 3 months in duration) (e.g., neck pain, thoracic pain, limb pain, low back pain) -OR-
* Chronic widespread pain (e.g., fibromyalgia, myofascial syndrome) -AND-
* 18 years of age or older -AND-
* Must be able to read, write, and speak English

Exclusion Criteria (as identified in referral package):

* Primary reason for referral stated as medication change or interventional pain management (e.g., injections, nerve block)
* Primary reason for referral is stated as headache or migraine.
* Reason for referral is chronic pelvic pain
* Referral includes information that patient has an untreated addiction, mental health disorder, or substance use disorder
* Referral indicates cancer-related pain
* Referral indicates medical "red flags" suggestive of non-musculoskeletal etiology of symptoms (e.g., unexplained symptoms, sudden weight loss, urinary retention, saddle anesthesia, evidence of upper motor neuron lesion, or fever)
* Referral states visceral pain or abdominal pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Participant recruitment | Baseline to 8 weeks
  Recruitment rate (participants/week) over 8 weeks.
Assessment completion | 12 months
  Proportion of all assessment items completed over the study duration (includes assessment items from baseline and 3, 6, 9, and 12 months follow-up)
Duration of baseline survey completion | Baseline
  Mean time to complete the baseline survey
Duration of follow-up survey completion | 12 months
  Mean time to complete follow-up surveys (includes surveys at 3, 6, 9, and 12 months)
Participant attrition | 12 months
  Attrition of participants expressed as a percentage lost to follow-up at 12 months.
Transfer of care | Baseline to 8 weeks
  Percentage of cases where the APP can successfully fulfill the role without having to transfer care to a physician or nurse practitioner as the most responsible provider.
Treatment fidelity | Baseline to 8 weeks
  Fidelity checklist for the APP intervention. Percentage of red flags screened for and percentage completion of all other assessment items.
Participant perspectives | 1-2 months after visit with APP
  Semi-structured interviews with participants involved in the study to explore acceptability of and satisfaction with the APP model of care.
Health care provider perspectives | 1-2 months after visit with APP
  Semi-structured interviews with health care providers involved in the study to explore acceptability of and satisfaction with the APP model of care.

SECONDARY OUTCOMES:
Brief Pain Inventory - pain severity subscale | Baseline and 3, 6, 9, and 12 months follow-up
  Numeric rating scale from 0 to 10, with higher scores indicating greater pain.
Brief Pain Inventory - pain interference subscale | Baseline and 3, 6, 9, and 12 months follow-up
  Numeric rating scale from 0 to 10, with higher scores indicating greater pain interference with 7 elements of daily living.
Health-related quality of life | Baseline and 3, 6, 9, and 12 months follow-up
  EuroQoL-5D-5L. This measure can be used in economic evaluations of health interventions. An index value is assigned and the EQ VAS is incorporated (0-100 scale, with higher scores representing better perceived health)
Pain Catastrophizing Scale | Baseline and 3, 6, 9, and 12 months follow-up
  Score of 0 to 52 with higher scores indicating greater catastrophic thinking.
Tampa Scale of Kinesiophobia | Baseline and 3, 6, 9, and 12 months follow-up
  17 items about pain-related fear. Higher scores (68 highest possible) suggesting worse pain-related fear.
Pain Self-Efficacy Questionnaire | Baseline and 3, 6, 9, and 12 months follow-up
  Score of 0 to 60, with higher scores suggesting higher confidence in dealing with pain.
Self-reported rating of change | 3, 6, 9, and 12 months follow-up
  Global rating of change scale of -5 to +5, with negative values showing a worsening of functional abilities and positive values an improvement in functional abilities.
Satisfaction with health care | 3, 6, 9, and 12 months follow-up
  Satisfaction with care will be assessed using an 11-point scale (-5 to +5). Negative scores demonstrate dissatisfaction and positive score suggest satisfaction with care.
Adverse events | 3, 6, 9, and 12 months follow-up
  Survey to ask participants if they experienced any adverse events related to treatment received. This includes the type of adverse event experienced, how long the event lasted, how bothersome the event was (0-10 scale), and what the participant thought caused the event.
Care provided | 12 months
  To describe the care provided, the investigators will present counts of following information from the participant's electronic medical records:
  * prescriptions for medications
  * assessments completed
  * interventions delivered
  * requisitions for diagnostic images
  * referrals to other health care providers
  * visits to other health care providers within the chronic pain clinic
  * notes to employers or insurers
Health utilization | 12 months
  From self-reported surveys, the investigators will collect the following health utilization measure counts related to the participant's chronic pain: emergency department visits, overnight hospitalizations, diagnostic images received, surgical interventions and pain injections/procedures, primary care visits (including walk-in clinic visits), specialist visits, medications used, other health care provider appointments (physiotherapy, occupational therapy, chiropractic, massage therapy, social worker visits, psychology), and self-care assistance required. These measures will be captured at 3, 6, 9, and 12 months to obtain cumulative measures and reduce the risk of recall bias. Note: medications will also be captured at baseline.
Health costs | 12 months
  Using the health utilization measures, cumulative direct healthcare costs (total costs and by health utilization measure) will be calculated using the Ontario Ministry of Health and Long-term Care Schedule of Benefits for publicly funded services and the Ontario Drug Benefit formulary for medication costs. For private services (e.g. PT in the community), the mean cost for the services in Kingston will be used.
Indirect costs | 12 months
  Indirect costs will be restricted to loss of productivity using a human capital approach. A dollar value will be assigned to time lost from paid employment (part-time, full-time, and self-employment) based on the mean wage in Ontario, according to Statistics Canada. The minimum wage in Ontario will be used to assign a value to time lost from volunteering, caregiving, or homemaking activities.

OTHER OUTCOMES:
Baseline measures | Baseline
  To describe the study population, the investigators will capture the following through the survey: age, gender, sex, education, identification as a member of a racialized group, identification as indigenous (First Nations, Inuit, Métis), duration and location of pain, current medications, work status, and annual household income.
Comorbidities | Baseline
  Self-Administered Comorbidity Questionnaire. Participants select relevant comorbidities from a list of specific problems (with three optional, open-ended conditions), whether they receive treatment for the condition, and whether the problem limits their activities.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Kingston Health Sciences Center, Hotel Dieu site - Chronic Pain Clinic, Kingston, Ontario
  - Queen's University, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.

REFERENCES:
- [Derived] Miller J, Doulas T, Bisson EJ, Abebe A, Chala M, McClintock C, Varette K, Vader K, Desmeules F, Perreault K, Donnelly C, Booth R, Tawiah AK, Duggan S. Assessing the feasibility of a clinical trial to evaluate an advanced practice physiotherapy model of care in chronic pain management: a feasibility study. Pilot Feasibility Stud. 2023 Jul 17;9(1):125. doi: 10.1186/s40814-023-01352-9. PMID 37461072